CLINICAL TRIAL: NCT04027244
Title: Leg Ischaemia Management Collaboration
Acronym: LIMb
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); National Institute for Health Research, United Kingdom (Other Government); The George Davies Charitable Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0686
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia; Frailty; Cognitive Impairment; Coronary Artery Disease
Keywords: Peripheral arterial disease; Limb salvage; Frailty; Cognitive dysfunction; Myocardial perfusion imaging; Biomarkers
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Frailty; Cognitive Dysfunction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Primary cohort: Any patient presenting to the Leicester Vascular Institute with SLI during the 2 year recruitment period (minimum 420 patients).
- Frailty & cognitive additional assessments: Any patient recruited to the primary cohort aged ≥65 years and undergoing an intervention for SLI (minimum 150 patients, target 210 patients).
- Cardiac MRI additional assessments: Any patient recruited to the primary cohort, with capacity to consent and undergoing an intervention for SLI (minimum 100 patients).
- Biomarkers additional assessments: Any patient recruited to the primary cohort and undergoing an intervention for SLI (no target recruitment set).
- Historical cohort: Retrospectively identified cohort of patients presenting to the study site with SLI between 2013 -15 (target 420).

SUMMARY:
Single-centre prospective cohort study of patients presenting with severe limb ischaemia (SLI). The primary outcome measure will be 12 month major amputation rate. A historical cohort of patients identified retrospectively will be the comparitor group used to assess the impact of a newly-established rapid-access limb salvage clinic.

Primary aim:

- Determine the proportion of patients with SLI undergoing major lower limb amputation within 12 months of presentation.

Secondary aims:

* Assess clinically important short-, medium- and long-term outcomes in those undergoing and not undergoing amputation
* Prevalence and degree of frailty and cognitive impairment
* Pevalence and degree of cardiac disease (detected by stress MRI)
* Establish a biobank for future biomarker analysis
* Investigate the role of frailty and cognitive assessments, cardiac MRI and biomarkers in risk-stratification of patients with SLI

DETAILED DESCRIPTION:
Severe limb ischaemia (SLI) is the end-stage of peripheral arterial occlusive disease (PAOD) whereby the viability of the limb is threatened due to the degree of arterial disease and subsequent ischaemia in the peripheral tissues. It is defined as ischaemic rest pain (or night pain) and/or ulceration or gangrene in the affected limb(s) for a minimum of two weeks attributed to confirmed PAOD. Treatment includes open surgical and endovascular revascularisation, with or without surgical debridement of affected tissues, amputation of toes and drainage of sepsis. In some patients revascularisation is not possible or fails resulting in the person requiring a major lower limb amputation.

Over 4000 major lower limb amputations per year were undertaken in England alone between 2003 and 2013 and a diabetes-related major lower limb amputation is performed every 30 seconds world-wide. As many as 25% of people with SLI will undergo a major lower limb amputation in the first year after presentation. Amputation negatively affects quality of life due to its negative impact on mobility, independence and ability to carry out activities of daily living.

This single-centre prospective cohort study will investigate the amputation rate at one year in patients presenting with SLI and compare this to a retrospectively identified historical cohort. This study will also investigate the prevelance and degree of frailty, cognitive impairment, and cardiac disease (detected by cardiac magnetic resonance imaging (MRI)), as well as establish a biobank for future biomarker analyses. The role of frailty and cognitive assessments, cardiac MRI and biomarker analysis in risk-stratifying patients with SLI will also be investigated.

ELIGIBILITY:
PRIMARY COHORT

Inclusion Criteria:

* All patients presenting to the Leicester Vascular Institute with SLI

Exclusion Criteria:

* SLI not caused by PAOD
* Patients undergoing intervention during their index presentation prior to recruitment
* Patients lacking capacity to consent with no accompanying next of kin, relative, partner or friend who can act as a personal consulted
* Patients who cannot read, write or understand English
* Any significant disease or disorder which may either put the patient at risk because of participation in the study, or may influence the results of the study or the patient's ability to participate in the study

FRAILTY & COGNITIVE ADDITIONAL ASSESSMENTS

Inclusion criteria:

* Patients recruited to the primary cohort in whom a decision has been made to undergo an intervention for SLI
* Patients aged ≥65 years

Exclusion criteria:

* Nil additional

CARDIAC MRI ADDITIONAL ASSESSMENTS

Inclusion criteria:

* Patients recruited to the primary cohort in whom a decision has been made to undergo an intervention

Exclusion criteria:

* Absolute contraindications to cardiac MRI (Pregnancy, Non-MR safe permanent pacemaker, implanted cardiac defibrillator, intra-auricular implant or intra-cranial clips, severe claustrophobia, unstable angina)
* Contraindication to gadolinium contrast agent (Known adverse reaction, chronic renal failure (eGFR <30mL/min/1.73m^2))
* Patients lacking capacity to consent for cardiac MRI

BIOMARKERS ADDITIONAL ASSESSMENTS

* Patients recruited to the primary cohort in whom a decision has been made to undergo an intervention

Exclusion criteria:

* Nil additional

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As representative a sample of patients presenting to the Leicester Vascular Institute with SLI during the study period as possible. All patients presenting with SLI within the age criteria will be eligible and personal consultee consent will allow recruitment even of those patients lacking capacity to consent.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-05-09 (Estimated); Study Completion 2031-05-09 (Estimated)

PRIMARY OUTCOMES:
12 month amputation rate | 12 months post recruitment
  Proportion of patients undergoing major lower limb amputation

SECONDARY OUTCOMES:
Amputation free survival | ≥12 months post recruitment
  Composite outcome measure of death or amputation
All-cause mortality | ≥12 months
  Death from any cause
Quality of life | 12 and 24 months post recruitment
  Quality of life as measured by the Vascular Quality of Life questionnaire (VascuQoL)
  * 25 item questionnaire, score 1-7 for each item, higher score = better quality of life
  * Domains: activities (8 items), symptoms (4 items), pain (4 items), social (2 items) and emotional (7 items); each scored 1-7 (total of domain item scores/number of items)
  * Overall score 1-7 (total item score/25)
Disability | 12 and 24 months post recruitment
  Level of disability as measured by the Barthel Index
  - Score 0-20; higher score = greater degree of functional independence/lower level of disability
Clinical Frailty Scale | Baseline, 12 and 24 months
  Prevalence and degree of frailty as measured by the Clinical Frailty Scale (CFS)
  * Score 1-9, higher score = greater degree of frailty
  * Results will also be reported dichotomised to frail (score ≥5) and non-frail (score ≤4)
Anxiety & Depression | Baseline, 12 and 24 months
  Prevalence and degree of anxiety and depression as measured by the Hospital Anxiety and Depression Scale (HADS)
  * 14 item questionnaire; score 0-3 for each item, higher score = more severe anxiety/depression
  * Domains: Depression (7 items), Anxiety (7 items); each scored 0-21; 0-7 = normal, 8-10 = bordeline, 11-21 = abnormal (case).

OTHER OUTCOMES:
Cognitive impairment (Frailty & Cognitive additional assessments only) | Baseline, 3 and 12 months
  Prevalence of cognitive impairment as detected by the Montreal Cognitive Assessment (MoCA)
  * Score 0-30; highger score = greater level of cognitive function
  * Results will also be reported dichotomised to normal (score ≥24) and cognitive impairment (score ≤23)
Post-operative delirium (Frailty & Cognitive additional assessments only) | 24 and 72 hours post intervention
  Incidence of post-operative delirium as detected by the Single Question in Delirium (SQiD) +/- 4 A's Test for delirium (4AT)
Prevalence of coronary artery disease (Cardiac MR additional assessments only) | Baseline
  Prevalence of coronary artery disease as detected by stress cardiac MRI
Incidence of peri-operative myocardial infarction (Cardiac MR additional assessments only) | 2-4 months post intervention
  Incidence of peri-operative myocardial infarction as detected by cardiac MRI
Edmonton Frail Scale (Frailty & Cognitive additional assessments only) | Baseline, 3 and 12 months
  Prevalence and degree of frailty as measured by the Edmonton Frail Scale (EFS)
  * Score 0-17, 0-5 = not frail, 6-7 = vulnerable, 8-9 = mild frailty, 10-11 = moderate frailty, 12-17 = severe frailty
  * Results will also be reported dichotomised to frail (score ≥8) and non-frail (score ≤7)

CONTACTS AND LOCATIONS:
Overall Officials: Rob D Sayers, MD, Study Chair — University of Leicester
Locations (1):
- Glenfield Hospital Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised dataset will be available on request to the Chief Investigator (Prof Rob Sayers). The study protocol will be published in an open-access journal prior to completion of recruitment.

REFERENCES:
- [Derived] Houghton JSM, Nduwayo S, Nickinson ATO, Payne TJ, Sterland S, Nath M, Gray LJ, McMahon GS, Rayt HS, Singh SJ, Robinson TG, Conroy SP, Haunton VJ, McCann GP, Bown MJ, Davies RSM, Sayers RD. Leg ischaemia management collaboration (LIMb): study protocol for a prospective cohort study at a single UK centre. BMJ Open. 2019 Sep 3;9(9):e031257. doi: 10.1136/bmjopen-2019-031257. PMID 31481569